CLINICAL TRIAL: NCT00970671
Title: Treatment of Surgical Scars With the 595nm Pulsed Dye Laser Using Purpuric and Nonpurpuric Parameters: A Comparative Study
Brief Title: Treatment of Surgical Scars Using the Pulsed Dye Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Julie Akiko Gladsjo, Clinical Instructor, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 090690
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Scar; Laser Therapy
Keywords: scar; laser therapy; lasers, pulsed dye
MeSH Terms: conditions — Cicatrix | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Laser treatment with Purpuric settings — Pulsed dye laser treatment at purpuric settings with pulse duration of 1.5msec.
  Other Names: Pulsed dye laser, 595nm VBeam, Candela
Other: Laser treatment with Nonpurpuric settings — Pulsed dye laser treatment with nonpurpuric settings with pulse duration 10msec.
  Other Names: Pulsed dye laser, 595nm VBeam, Candela
Other: No treatment — No laser treatment

SUMMARY:
The purpose of this study is to determine whether treatment of fresh surgical scars with a pulsed dye laser using purpura-inducing settings will improve clinical appearance better than one using non-purpura-inducing settings or no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring Mohs micrographic surgery or excisions for skin cancer or atypical nevi, with an expected post-excision scar of 4.5cm in length or more.
* Willing to participate.
* Able to give informed consent

Exclusion Criteria:

* Location of excision or Mohs surgery on the genitals, hands, or feet.
* Fitzpatrick skin type V or VI.
* Prior history of known light sensitivity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale score | 6weeks, 10weeks, and 18weeks after surgery

SECONDARY OUTCOMES:
Subjective rating of pain on scale of 0 to 10 | at each treatment visit: 2weeks, 6weeks, and 10weeks after surgery
Cosmetic appearance of scar | 6weeks, 10 weeks, and 18weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Gladsjo, MD PhD, Principal Investigator — University of California, San Diego; S. Brian Jiang, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Perlman Ambulatory Center - Dermatology clinic, La Jolla, California, United States